CLINICAL TRIAL: NCT05456633
Title: Multi-Center, Retrospective and Prospective Evaluation for Clinical and Radiographic Outcomes of Spine Surgeries Utilizing Capri Cervical and Thoracolumbar Corpectomy Cage Systems: Observational Post Market Clinical Follow-Up Study
Brief Title: Clinical and Radiographic Outcomes of Spine Surgeries Utilizing Capri Cervical and Thoracolumbar Corpectomy Cage Systems
Status: Withdrawn | Type: Observational
Why Stopped: The study has been withdrawn and no participant was enrolled.
Sponsor: K2M, Inc. (Industry)
Collaborators: Stryker Spine (Industry)
Responsible Party: Sponsor
Other Study IDs: CAS-031
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Thoracolumbar Spine; Cervical Spine Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Capri Cervical 3D Static: Subjects who have undergone or will undergo VBR in the cervical spine (C2 to T1 in the USA, C3 to C7 outside of the USA) to replace diseased or damaged vertebral bodies due to tumor, trauma (i.e., fracture), or osteomyelitis, or for reconstruction following corpectomy performed to achieve decompression of the spine cord and neural tissues in cervical degenerative disorders
  Interventions: Device: Capri Cervical Static
- Capri Cervical 3D Expendable: Subjects who have undergone or will undergo VBR in the cervical spine (C2 to T1 in the USA, C3 to C7 outside of the USA) to replace diseased or damaged vertebral bodies due to tumor, trauma (i.e., fracture), or osteomyelitis, or for reconstruction following corpectomy performed to achieve decompression of the spine cord and neural tissues in cervical degenerative disorders
  Interventions: Other: CAPRI Static Expandable
- Capri Thoracolumbar Expandable: Subjects who have undergone or will undergo VBR in the thoracolumbar spine (T1 to L5) with Capri Thoracolumbar Expandable to replace collapsed, damaged, or unstable vertebral bodies due to tumor or trauma (i.e., fracture)
  Interventions: Device: Capri Thoracolumbar

INTERVENTIONS:
Device: Capri Cervical Static — When used in the cervical spine (C2-T1), CAPRI Static cages are intended for use in skeletally mature patients to replace a diseased or damaged vertebral body caused by tumor, fracture, or osteomyelitis, or for reconstruction following corpectomy performed to achieve decompression of the spinal cord and neural tissues in cervical degenerative disorders.
  Groups: Capri Cervical 3D Static
Other: CAPRI Static Expandable — When used in the cervical spine (C2-T1), CAPRI Static Expandable cages are intended for use in skeletally mature patients to replace a diseased or damaged vertebral body caused by tumor, fracture, or osteomyelitis, or for reconstruction following corpectomy performed to achieve decompression of the spinal cord and neural tissues in cervical degenerative disorders.
  Groups: Capri Cervical 3D Expendable
Device: Capri Thoracolumbar — Intended for use to replace a collapsed, damaged, or unstable vertebral body due to tumor and trauma (i.e. fracture).
  Groups: Capri Thoracolumbar Expandable

SUMMARY:
This is a retrospective and prospective observational, multi center study of subjects who have undergone or will undergo vertebral body replacement surgery in the cervical or thoracolumbar spine utilizing Stryker Capri Corpectomy Cages.

The primary study hypothesis to determine effectiveness, is that the mean improvement in NDI (cervical) or ODI (thoracolumbar) score from baseline meets or exceeds 15-points at 24 months for Stryker Capri Corpectomy Cage systems individually.

DETAILED DESCRIPTION:
Corpectomy procedures are utilized to treat a variety of spinal pathologies including tumor, often as a result of metastatic spine disease, fracture frequently attributed to trauma, osteomyelitis (infection), and degenerative disorders which require reconstruction to achieve decompression of the spinal cord or neural tissues. Patients may present with pain, spinal instability, and neurological deficits. Corpectomy involves a resection or excision of the affected vertebrae and intervertebral disc(s), followed by placement of a vertebral body replacement (VBR) to reconstruct the anterior column of the spine and restore stability and alignment.

Common indications for VBR procedures include spinal instability due to vertebral fractures, vertebral compression fractures, and fractures related to malignancy or infection and control of disease, such as metastatic disease in the spine. Causes of spinal fractures may include falls, sports, and motor vehicle accidents. Spinal tumors are often caused by metastases of the skeletal system, which commonly affect the spine. Additionally, VBR procedures may be considered in response to cervical spondylotic myelopathy which is a progressive degenerative disease and a common cause of cervical spinal cord dysfunction and cervical myelopathy in people over the age of 55. Corpectomy (or vertebrectomy) with reconstruction has become a common surgical procedure used for decompression and reconstruction of the spine. Traditionally, reconstruction has included autograft, allograft, and bone substitutes; however, the use of grafts alone have been reported to lead to complications such as donor site morbidity, high rates of pseudarthrosis, and delayed union. The evolution of corpectomy cages has led to improvements in both clinical and radiographic outcomes. Titanium mesh cages were one of the earliest types of non-graft-based corpectomy cages, providing a biocompatible method of rapidly stabilizing the affected segments, reducing donor site morbidity, and improving outcomes.

This study will examine use of the Capri Corpectomy Cage systems in cervical and/or thoracolumbar cases in the treatment of trauma, tumor, infection (cervical only), or degeneration (cervical only) using static (cervical only) or expandable (cervical and thoracolumbar) cages. Clinical efficacy and safety will be assessed in this post-market study through evaluation of patient outcomes in comparison to baseline, pre-operative conditions.

Capri Corpectomy system implants are VBR devices that are designed in a variety of lengths, widths, and heights to match the patient's anatomy. The caudal and cephalad ends of the implant have teeth which are designed to engage with the vertebral body endplates. The side walls of the implants contain windows that may be used for graft incorporation. Instruments are used for inserting the associated implant components using standard surgical techniques. There are curettes, scrapers, and box chisels for preparing the disc spaces and vertebral body endplates. Insertion instruments are available for inserting the implant. Capri Corpectomy Cage systems are available as cervical static cages (comprised of titanium alloy) and cervical or thoracolumbar adjustable (i.e., expandable) cages (comprised of titanium alloy and cobalt chrome). Devices may be implanted via posterior, anterior, or lateral approaches.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature
* Willingness and ability to comply with the requirements of the protocol including follow-up requirements
* Willing and able to sign a study specific informed consent form. For fully retrospective enrollments, i.e., subjects that already have 24-month follow-up data available, the Principal Investigator will request a waiver of the written informed consent requirement.
* Has undergone or will undergo VBR in the cervical spine (C2 to T1 in the USA, C3 to C7 outside of the USA) using either Capri Cervical 3D Static OR Capri Cervical 3D Expandable to replace diseased or damaged vertebral bodies due to tumor, trauma (i.e., fracture), or osteomyelitis, or for reconstruction following corpectomy performed to achieve decompression of the spine cord and neural tissues in cervical degenerative disorders -OR- Has undergone or will undergo VBR in the thoracolumbar spine (T1 to L5) using Capri Thoracolumbar Expandable to replace collapsed, damaged, or unstable vertebral bodies due to tumor or trauma (i.e., fracture)
* Score at least 30 points on the ODI or at least 30 points on the NDI at screening (or before surgery for retrospective enrollment) (on a 100-point scale)

Exclusion Criteria:

* Presence of infection, except within the spinal indications for use of this product
* Pregnancy (pregnant at the time of enrollment or intends to become pregnant during the course of the study)
* Metabolic disorders of calcified tissues
* Grossly distorted anatomy
* Inadequate tissue coverage
* Drug / alcohol abuse
* Mental illness such as a psychiatric or cognitive impairment, that in the opinion of the investigator, would interfere with the subject's ability to comply with the study requirements or patient reported outcomes (e.g., Alzheimer's Disease)
* General neurological conditions
* Immunosuppressive disorders
* Subjects with known sensitivities to materials in the device
* Obesity defined as a BMI greater than 30
* Subjects who are unwilling to restrict activities or follow medical advice
* Any condition where the implants interfere with anatomical structures or precludes the benefit of spinal surgery
* Biological factors such as smoking, use of nonsteroidal anti-inflammatory agents, use of anticoagulants, etc.

  * Subjects that adhere to the specified washout period detailed below can be enrolled: Smoking cessation must occur at a minimum of 4 weeks prior to surgery; Nonsteroidal anti-inflammatories (NSAIDs) should be stopped at a minimum of 7 days prior to surgery; Anticoagulants should be stopped at the discretion of the operating surgeon as the washout period varies for each medication
  * Trauma subjects that are unable to adhere to the washout period can be enrolled; however, the aforementioned biological factors will need to be documented during data collection
* Prior fusion at the level(s) to be treated
* Incarcerated at the time of study enrollment
* Current participation in an investigational study that may impact study outcomes
* Involved in current or pending spinal litigation or a workman compensation claim

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The sample size for this study will be a total of 126 subjects planned to receive one of the Capri Corpectomy systems mentioned below at up to 20 sites in the United State:
  * 42 subjects for Capri Cervical 3D Static
  * 42 subjects for Capri Cervical 3D Expandable
  * 42 subjects for Capri Thoracolumbar Expandable This sample size allows for up to a 15% loss-to-follow-up at 24 months. The sample size analysis below indicates that N=36 per device are needed for 80% power to meet the a priori performance goal
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mean improvement in NDI score | 24 Months
  Mean improvement in NDI score over baseline that meets or exceeds 15 points (on a 100 point scale) at 24 months (cervical)
Mean ODI improvement | 24 Months
  Mean ODI improvement over baseline that meets or exceeds 15 points (on a 100-point scale) at 24 months (thoracolumbar)

SECONDARY OUTCOMES:
NDI or ODI | Initial Post-Op to 24 Months
  Patient-Reported Outcome Measures
Visual Analogue Scale (VAS) | Initial Post-Op to 24 Months
  Patient-Reported Outcome Measures
EuroQol-5 Dimensions-5 Levels (EQ 5D-5L) | Initial Post-Op to 24 Months
  Patient-Reported Outcome Measures
Fusion or non-union | 24 Months
  Radiographic Assessments: Effectiveness
Range of motion | 24 Months
  Radiographic Assessments: Effectiveness
Translational motion | 24 Months
  Radiographic Assessments: Effectiveness
Disc height | 24 Months
  Radiographic Assessments: Effectiveness
Surgery Time | During Surgery
  Clinical Observations
Anesthesia Time | During Surgery
  Clinical Observations
Estimated blood loss | During Surgery
  Clinical Observations
Length of hospital stay on day of Surgery / Pre-Discharge | During Surgery
  Clinical Observations
Patient Satisfaction at 12 Month | 12 Months
  Clinical Observations
Patient Satisfaction | 24 Months
  Clinical Observations
Use of pain medication post surgery at all visits | Post surgery - 24 Months
  Clinical Observations
Neurological Examination | 12 Months
  Clinical Observations
Subsidence | 12 and 24 Months
  X-Ray Safety Assessment
Device Migration | 12 and 24 Months
  X-Ray Safety Assessment
Adjacent Segment Degeneration | 12 and 24 Months
  X-Ray Safety Assessment
Device and supplemental fixation breakage | 12 and 24 Months
  X-Ray Safety Assessment